CLINICAL TRIAL: NCT04303117
Title: Phase I/II Study of PDS01ADC Monotherapy and in Combination With M7824 in Advanced Kaposi Sarcoma
Brief Title: NHS-IL12 Monotherapy and in Combination With M7824 in Advanced Kaposi Sarcoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 200061; 20-C-0061
Record Dates: First submitted 2020-03-07; First posted 2020-03-10 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08-20

CONDITIONS: Kaposi Sarcoma
Keywords: Immune Therapy; AIDS; HIV; Immunocytokine
MeSH Terms: conditions — Sarcoma, Kaposi; Acquired Immunodeficiency Syndrome | interventions — NHS-IL12 immunocytokine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1/Monotherapy (Experimental): Treatment with NHS-IL12 at de-escalating doses if necessary
  Interventions: Drug: NHS-IL12
- Arm 1a/Monotherapy Expansion (Experimental): Treatment with NHS-IL12 at MTD
  Interventions: Drug: NHS-IL12
- Arm 2/Combination therapy (Experimental): Treatment with NHS-IL12 at MTD and M7824 at a fixed dose
  Interventions: Drug: NHS-IL12; Drug: M7824

INTERVENTIONS:
Drug: NHS-IL12 — An initial dose of 16.8 mcg/kg administered subcutaneously every 4 weeks and at an MTD dose with M7824 on day 1 of a 28-day cycle.
Drug: M7824 — 1200 mg administered IV every two weeks while on NHS-IL12.
  Arms: Arm 2/Combination therapy

SUMMARY:
Background:

Kaposi sarcoma (KS) tumors grow on the skin, lymph nodes, lungs, bone, and gastrointestinal tract. KS often affects people with immune deficiencies, such as among people living with HIV or those with prior history of transplant. Researchers want to see if 2 non-chemotherapy drugs can help people with KS. NHS-IL12 triggers the immune system to fight tumors. M7824 blocks the pathways that cancer cells use to stop the immune system from fighting tumors.

Objective:

To learn if giving NHS-IL12 alone or with M7824 could help the immune system fight KS tumors.

Eligibility:

People 18 and older with KS that has been treated with chemotherapy or immunotherapy

Design:

Participants will be screened with some or all of the following:

medical history

physical exam

chest X-ray

computed tomography scan

blood and urine tests

electrocardiogram and echocardiogram

skin KS lesion biopsy

lung exam

gastrointestinal exam

All participants will get NHS-IL12 every 4 weeks for up to 96 weeks (or 24cycles). It is injected under the skin.

Some participants will also get M7824 every 2 weeks for up to 96 weeks (or 24cycles). It is given through a plastic tube that is put in an arm vein.

Participants will complete questionnaires about how KS affects their quality of life. Their KS lesions will be measured and photographed. They will repeat some of the screening tests. They will give saliva samples or additional tissue samples. They will have a lung function test. Their ability to perform their normal activities will be assessed. The treatment duration is up to 96 weeks (or 24cycles) with an option to take NHS-IL12 and/or M7824 until the KS tumors are not responding, or you develop unacceptable side effects.

Participants will have follow-up visits 7 and 30 days after treatment ends, then every 3 to 6 months for the next 18 months, then once a year for 3 years.

DETAILED DESCRIPTION:
Background:

* Kaposi Sarcoma (KS) is a multicentric angioproliferative tumor, caused by Kaposi sarcoma-associated herpesvirus, that most frequently involves the skin, but may also involve lymph nodes, lungs, bone and gastrointestinal tract. It is most common in people with HIV but may also occur in patients without a diagnosis of HIV. Patients with HIV-associated KS have worse survival than HIV-infected patients without KS.
* As it is a relapsing and remitting condition, patients with KS often require prolonged courses of cytotoxic chemotherapy.
* KS is an immune responsive tumor as interferon-alpha, pomalidomide, and restoring T-cell function in HIV + patients treated with antiretroviral drugs can result in clinical benefit and remission of KS.
* Published Phase I/II studies by our group demonstrated that IL-12 alone and in combination with liposomal doxorubicin led to clinical responses in patients with advanced KS.
* PDS01ADC is an immunocytokine with affinity to both single and double stranded DNA allowing for targeting of exposed DNA, which is commonly seen in necrotic tumors. This agent is able to deliver IL-12 to the tumor microenvironment promoting local immunomodulation, that results in less systemic toxicity than IL-12 systemic administration.
* M7824 is a novel bifunctional fusion protein composed of a monoclonal antibody against human PD-L1 (avelumab) fused with the extracellular domain of human TGF-beta receptor II (TGF-betaRII), which functions as a TGF-beta trap .
* Anti-PD-L1 and anti-PD-1 agents have been found to be active in certain virus-induced cancers, including Kaposi sarcoma, and to be safe and active in patients with HIV infection.
* Currently, no clinical data exists for the combination of PDS01ADC and M7824. Preclinical data suggest synergy between these agents from existing ongoing studies and the available clinical data both in KS and other tumor subtypes suggest that the combination of PDS01ADC with M7824 is likely to be well-tolerated and has scientific rationale. This combination offers a new treatment approach for patients with advanced KS who have received prior therapies.

Objectives:

-Evaluate the safety, tolerability, and activity of single agent PDS01ADC and the combination of PDS01ADC with M7824 in participants with advanced KS

Eligibility:

* Age >=18 years
* Histologically confirmed Kaposi sarcoma (KS)
* KS requiring systemic therapy, with or without a history of prior systemic therapy
* At least five measurable cutaneous KS lesions with no previous local radiation, surgical or intralesional cytotoxic therapy to these measurable lesions.
* ECOG Performance Status (PS) <= 2
* Participant must be willing to give informed consent.
* Participants can be HIV positive or negative.
* Antiretroviral therapy (ART) for HIV+ participants for 8 or more weeks prior to entry with an HIV viral load of <400 copies/ml and CD4+ T-cell count >50 cells/microliter.
* Participants with bleeding from visceral sites of KS or requiring blood transfusions in the 2 weeks prior to study entry will not be eligible.

Design:

* This is a Phase I/II study assessing the safety and efficacy of PDS01ADC alone or in combination with M7824 in participants with advanced KS. Participants will receive therapy until optimal tumor response, unacceptable toxicity, the participant s request to discontinue therapy, PI decision, up to a total of 96 weeks, or 24 cycles.
* Monotherapy: Participants with history of prior systemic therapy will receive PDS01ADC alone with a 3+3 design applicable to the first 3-6 participants at a starting dose of 16.8 microgram/kg on day 1 of a 28-day cycle. Two dose de-escalation levels (Dose Level -1: 12 microgram/kg or Dose Level -2: 8 microgram/kg) will be permitted if there is evidence of 2 or more dose limiting toxicities within the first 6 weeks of therapy. An expansion cohort will investigate the activity of PDS01ADC in participants with and without prior systemic therapy for KS.
* Combination Therapy: The combination arm will open following accrual and completion of the DLT period for participants in the monotherapy arm. Up to 28 participants will be treated with M7824 (1200 mg IV, every 2 weeks) and PDS01ADC (MTD dose from the monotherapy arm). The DLT period for this arm will be 6 weeks.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Individuals with biopsy proven (confirmed in the Laboratory of Pathology, CCR) Kaposi sarcoma (KS)
* KS requiring systemic therapy, with or without history of prior KS therapy:

  * T1 KS or T0 KS sufficiently widespread that systemic therapy is advisable, or KS affecting quality-of-life due to local symptoms or psychological distress

OR,

* KS with an inadequate response to liposomal doxorubicin, paclitaxel, other systemic chemotherapy (either progressive disease or stable disease after 3 or more cycles) or immunotherapy (progressive disease)

  * A wash-out period off treatment of 2 weeks from last chemotherapy and 4 weeks from last immunotherapy, other systemic treatment with a biologic agent, or monoclonal antibody therapy will be required in individuals with prior KS therapy.
  * Resolution of toxicity from prior therapy to <= Grade 1.
  * At least five measurable cutaneous KS lesions with no previous local radiation, surgical or intralesional cytotoxic therapy that would prevent response assessment for that lesion.
  * Measurable disease by the criteria proposed by the AIDS Clinical Trials Group (ACTG) Oncology Committee for KS
  * HIV positive or negative.
  * ART for HIV+ individuals for 8 or more weeks prior to entry with an HIV viral load of <400 copies/ml at screening and CD4+ T cell count of >= 50 cells/microliter as this may be expected if individuals have received several courses of chemotherapy.
  * Age >=18 years.
  * ECOG performance status <=2 (Karnofsky >=60%).
  * Adequate organ and marrow function as defined below:
* Absolute neutrophil count >=1,000/mcL
* Platelets >=100,000/mcL
* Total bilirubin within normal institutional limits; OR <3x institutional ULN for Gilbert s syndrome or HIV protease inhibitors; OR <5x ULN and direct bilirubin < 0.7mg/dL for individuals on atazanavir-containing HIV regimen
* AST(SGOT)/ALT(SGPT) <=1.5 X institutional upper limit of normal
* Hemoglobin >= 9g/dL
* Creatinine within normal institutional limits OR creatinine clearance >30 mL/min/1.73m^2 as estimated by either Cockroft-Gault of 24- hour urine collection if creatinine levels above institutional normal

  * Normal international normalized ratio (INR), PT<=1.5 x ULN and activated partial thromboplastin time (aPTT) <= 1.5 x ULN
  * The effects of PDS01ADC and M7824 on the developing human fetus are unknown. For this reason, individuals of child-bearing potential (IOCBP) and individuals able to father a child must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, during treatment and for at least 4 months after the last dose of treatment and agree to inform the treating physician immediately if they become pregnant. Also, there is unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with M7824 and/or PDS01ADC, therefore IOCBP must agree to discontinue nursing if treated with these agents.
  * Ability of individual to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Receiving any other investigational agents.
* Pregnant individuals are excluded from this study as the effects of PDS01ADC and M7824 have potential teratogenic or abortifacient effects.
* Severe KS (such as symptomatic pulmonary KS) that could be life threatening if it progressed over 2-4 weeks
* Actively bleeding sites caused by visceral KS.
* Unwilling to accept blood products as medically indicated
* Actively bleeding and/or requiring transfusions in the 2 weeks preceding study entry.
* History of bleeding, diathesis, or recent major bleeding events within a period of 4 weeks considered by the investigator as high risk for investigational drug treatment.
* Any active or recent history (symptomatic in the last 3 months) of a known or suspected autoimmune disease (with the exception of diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment) or recent history of a syndrome that required systemic corticosteroids (10mg daily prednisone or equivalent) or immunosuppressive medications except inhaled steroids and adrenal replacement steroids doses up to 10mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Uncontrolled opportunistic infections
* Active multicentric Castleman disease
* Individuals with primary effusion lymphoma
* History of malignant tumors other than KS, unless:

  * In complete remission for >= 3 years from the time complete remission was first documented or
  * Resected basal cell or squamous cell carcinoma of the skin or
  * In situ cervical or anal dysplasia
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to PDS01ADC and/or M7824 investigational agents used in study.
* Active tuberculosis (TB):

  * Individuals who are undergoing first month of therapy (RIPE or equivalent) for active TB or
  * Individuals with TB immune reconstitution syndrome (IRIS) requiring corticosteroids
* Received or will receive a live vaccine within 30 days prior to the first administration of study intervention. Seasonal flu vaccines that do not contain a live virus are permitted. Locally approved COVID vaccines are permitted.
* Uncontrolled substantial intercurrent illness including, but not limited to, ongoing or active severe infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, that would limit compliance with study requirements.
* Medical or psychiatric illness or social situation that would, in the opinion of the investigator, preclude participation in the study or the ability of individuals to provide informed consent for themselves.
* Uncontrolled HBV infection, defined as plasma HBV DNA detectable by PCR

Note: the following will NOT be exclusionary:

* A positive hepatitis B serology indicative of previous immunization (i.e. HbsAb positive and HbcAb negative), or a fully resolved acute HBV infection
* Chronic HBV suppressed by appropriate antiretroviral therapy with activity against HBV, as outlined in DHHS guidelines.

  * Uncontrolled HCV infection, defined as plasma HCV DNA detectable by PCR

Note: the following will NOT be exclusionary:

* Positive HCV serology but no detectable HCV RNA, indicative of spontaneously cleared HCV infection
* Successfully treated for HCV as long as therapy for HCV has been completed.

  -Individuals will be excluded from the combination therapy arm if:
* they have discontinued prior PD1/L1 blocking agent due to immune mediated adverse event(s) OR
* they have active non-infectious pneumonitis or a history of steroid requiring non-infectious pneumonitis.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-07-13 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
safety, tolerability and activity of NHS-IL12 alone or in combination with M7824 | 24 cycles of treatment, until confirmed progression, unacceptable toxicity or trial withdrawal
  The fraction of participants with toxicity noted at each dose level will be reported by grade and type of toxicity identified. Maximum tolerated dose will also be reported.

SECONDARY OUTCOMES:
progression free survival | every 3 months for the first 6 months after completion of therapy, then every six months for the next 18 months, and then annually for a total of 3 years
  duration of time from the start of the treatment until time of disease relapse from PR, disease progression, or death, whichever occurs first
objective response rates | every 3 months for the first 6 months after completion of therapy, then every six months for the next 18 months, and then annually for a total of 3 years
  Percentage of participants with the best overall response of CR or PR to therapy
duration of response | every 3 months for the first 6 months after completion of therapy, then every six months for the next 18 months, and then annually for a total of 3 years
  the time criteria are met for CR or PR (whichever is recorded first) until the first date that participant no longer qualifies as a PR

CONTACTS AND LOCATIONS:
Overall Officials: Ramya M Ramaswami, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-C-0061.html